CLINICAL TRIAL: NCT06889779
Title: A Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy of Two Different Mixes of HMO-2FL + Humiome® Post LB Postbiotic (Postbiotic-LB) on Gastrointestinal Symptoms in Irritable Bowel Syndrome (IBS) Subjects
Brief Title: Study Evaluating the Efficacy of Different Mixes of HMO-2FL + Humiome® Post LB on IBS Gastrointestinal Symptoms
Acronym: DORPHI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-08-14-DORP
Record Dates: First submitted 2025-02-20; First posted 2025-03-21 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-02

CONDITIONS: IBS (Irritable Bowel Syndrome)
Keywords: Dietary supplement IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel Assignment A randomized, placebo-controlled, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MIX 1 (Active Comparator): Humiome® Post LB postbiotic 300 mg , Human Milk Oligosaccharides 2'-O-fucosyllactose 300 mg 1 capsule per day orally
  Interventions: Dietary Supplement: MIX 1
- MIX 2 (Active Comparator): Humiome® Post LB postbiotic 100 mg Human Milk Oligosaccharides 2'-O-fucosyllactose 500 mg 1 capsule per day orally
  Interventions: Dietary Supplement: MIX 2
- Placebo (Placebo Comparator): Microcrystalline 1 capsule per day orally
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MIX 1 — Humiome® Post LB postbiotic 300 mg , Human Milk Oligosaccharides 2'-Ofucosyllactose 300 mg 1 capsule per day Orally
  Arms: MIX 1
Dietary Supplement: MIX 2 — Humiome® Post LB postbiotic 100 mg Human Milk Oligosaccharides 2'-O-fucosyllactose 500 mg 1 capsule per day Orally
  Arms: MIX 2
Dietary Supplement: Placebo — Microcrystalline cellulose 1 capsule per day Orally
  Arms: Placebo

SUMMARY:
A randomized, placebo-controlled, double-blind clinical study to evaluate the efficacy of two different mixes of HMO-2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB) on Gastrointestinal Symptoms in individuals with Irritable Bowel Syndrome (IBS)

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, double-blind clinical trial designed to assess the efficacy of two distinct formulations combining Human Milk Oligosaccharide 2'-O-fucosyllactose (HMO-2FL) with Humiome® Post LB postbiotic (postbiotic-LB) in alleviating gastrointestinal symptoms in individuals with Irritable Bowel Syndrome (IBS). Participants will be randomly assigned to receive either of the two active formulations or a placebo, ensuring unbiased comparisons. We aim to evaluate changes in gastrointestinal symptoms, including abdominal pain, bloating, and bowel movement patterns, using validated symptom scoring tools. We will assess the quality of life, gut health biomarkers, and safety profiles. The study employs a double-blind design, where neither participants nor investigators will know the treatment assignments, maintaining the study's integrity. By comparing the effects of different HMO-2FL and postbiotic-LB combinations, this trial aims to provide evidence-based insights into novel dietary supplement options for IBS management, contributing to the growing field of gut health and microbiome-targeted solutions.

ELIGIBILITY:
* Written and signed informed consent (will be obtained before any study-related Assessments).
* Male or female aged ≥18 - 70 years at the time of consent.
* Female individuals of childbearing potential (Females who are peri or post-menopausal, i.e., when there has been no or irregular menstruation for a minimum of 12 months prior to screening, are considered not to be of child-bearing potential.), who are not surgically sterilized, must have a negative pregnancy test at screening and be willing to practice one of the following appropriate contraceptive methods until:

  * Sexual abstinence.
  * Oral contraceptives.
  * Trans-dermal patches or depot
  * injection of a progestogen drug (starting at least 4 weeks prior to product administration).
  * Double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent.
  * Intrauterine device (IUD), intrauterine system (IUS), subdermal implant, or vaginal ring (placed at least 4 weeks prior to product administration/2 weeks prior screening).
  * Contraceptives must be effective before the randomization visit.
* Individuals with plasma FBG (fasting blood glucose) (less than equal to 125 mg/dl).
* Individuals with Hemoglobin (Hb%) (more than equal to 10 g/dl).
* Individuals with BP (blood pressure) (less than equal to 140/100 mm Hg)
* Individuals with normal haematology as assessed by CBC (complete blood counts)
* Individuals with TSH levels in between 0.4 mIU/L to 5.0 mIU/L
* Individuals with SGOT and SGPT within 2 X the Upper normal limit (ULN) and serum
* Individuals with creatinine within 1.5 X ULN
* Rome-IV diagnostic criteria: Individuals with more than 25% of bowel movements with Bristol stool types 1, 2 or 6,7 and have had recurrent abdominal pain, on average, at least 1 day/week in the last 3 months. And the pain is associated with two or more of the following criteria:

  * Related to defecation
  * Associated with a change in frequency of stool
  * Associated with a change in form or appearance of stool as
  * assessed by Bristol stool types 1,2, 6 or 7.
  * Individuals meeting the above criteria for the last 3 months with
  * symptom onset at least 6 months before diagnosis
* Individuals with Abdominal pain severity (more than equal to 6 on a 11-point scale) at screening and during placebo run-in period.
* Individuals with IBS-SSS of at least 175 points at screening.
* Individuals who are mentally stable as assessed by Perceived Stress Scale (PSS) less than equal to 26 (Low to Moderate stress).
* Individuals who understand the nature and purpose of the study including the potential risks and side effects.
* Individuals who are willing to complete all study procedures including study-related questionnaires and comply with study requirements.
* Individuals who are capable of filling the app-based digital form/diary.

Exclusion Criteria:

* Individuals with IBS-M.
* Treatment with an investigational drug within 30 days/5 half-lives of the drug (whichever longest) prior to screening visit.
* Individuals with organic disease like infectious diseases, inflammatory diseases, metabolic disorders, neurological diseases, autoimmune disorders, cancer etc. (to be ruled out by physician based on prior history and physical examination).
* Individuals with a history of surgical resection of the stomach, small intestine or large intestine.
* Individuals with a history of or complications from inflammatory bowel disease (Crohn's disease or ulcerative colitis), colitis and enteritis.
* Individuals with a history of any diet-based intolerance (gluten or lactose intolerance).
* Individuals with a history of drug or alcohol abuse within the past 6 months.
* Individuals with severe depression or an anxiety disorder, which could potentially affect the efficacy evaluation (as determined by the qualified investigator).
* Individuals with uncontrolled hypertension or on antihypertensive medications.
* Individuals with serious cardiovascular diseases, respiratory diseases, renal diseases, hepatic diseases, gastrointestinal diseases (excluding IBS), blood diseases or neurological or psychiatric diseases.
* Individuals who are pregnant, breastfeeding or planning on becoming pregnant throughout the course of the study.
* Individuals with Type I or Type II diabetes mellitus.
* Individuals with a history of or current diagnosis of any cancer diagnosed less than 5 years prior to screening. Individuals with cancer in full remission more than 5 years after diagnosis are acceptable.
* Individuals who are immuno-compromised (HIV positive, on antirejection medication, rheumatoid arthritis and other autoimmune disorders).
* Individuals with a history of abdominal surgery.
* Individuals with diarrhoea of any other origin.
* Individuals currently or in future planning to fast for more than 24 hours.
* Individuals with an active eating disorder.
* Individuals who have used an over-the-counter or prescription laxative medication or any other herbal agents affecting GI motility within 2 weeks prior to screening.
* Individuals who have used pre/pro/post/synbiotic, Human Milk Oligosaccharides (HMOs), or fiber supplements (or probiotic/fiber enriched foods) or FODMAP diet or an antibiotic within 4 weeks prior to screening.
* Individuals who have used IBS specific treatments within 4 weeks prior to screening.
* Individuals who currently consume greater than 2 standard alcoholic drinks per day from past 3 months. ((One unit of alcohol is equal to 45 ml of hard liquor, 150 ml of wine or a pint of beer)
* Smokers (in any number and any format)
* Individuals with an allergy or sensitivity to the probiotic products.
* Individuals who are cognitively impaired and/or who are unable to give an informed consent.
* Individuals who have abnormal laboratory results or any other medical or psychological condition which, in the opinion of the qualified investigator, may adversely affect the Individuals' ability to complete the study or its measures or which may pose significant risk to the individual.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB) on IBS symptoms as assessed by IBS Symptom Severity Scale (IBS-SSS), when compared to placebo | Day 0 & Day 42
  The IBS Severity Scoring System (IBS-SSS) will be used to assess symptom severity. Participants will rate their symptoms over the last 10 days on day 0 and day 42. The change in the average IBS severity score will be calculated and compared to the placebo group.

SECONDARY OUTCOMES:
To assess the efficacy of daily consumption of two different mixes of HMO 2'-O-fucosyllactose + Humiome® Post LB postbiotic on IBS symptoms as assessed by IBS Symptom Severity Scale , when compared to placebo in individuals | Day 0, Day 21
  The IBS Severity Scoring System (IBS-SSS) will be used to assess symptom severity. Participants will rate their symptoms over the last 10 days on day 0 and day 21. The change in the average IBS severity score will be calculated and compared to the placebo group.
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on IBS symptoms as assessed by IBS-SSS, when compared to baseline in individuals with IBS | Day 0, Day 21 and Day 42
  The IBS Severity Scoring System (IBS-SSS) will be used to assess symptom severity. Participants will rate their symptoms over the last 10 days on day 0 and day 42. The change in the average IBS severity score will be calculated and compared to baseline in individuals with IBS.
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on Abdominal Pain severity compared to baseline, each other and placebo in individuals with | Day 0, Day 21 and Day 42
  Decrease in Abdominal pain severity as assessed by APS-NRS (Abdominal pain severity - Numeric rating scale)
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose + Humiome® Post LB postbiotic on participant by Stool consistency (Bristol Stool Form Scale types 3, 4 & 5) | Time Frame: Day 0, Day 21 and Day 42
  In gastroenterology, stool consistency is commonly measured using the Bristol Stool Form Scale (BSFS), which categorizes stool into seven types, from type 1 (hard lumps) to type 7 (watery diarrhea). It is a simple, cost-effective tool used as a marker for intestinal transit time and bowel function. In this study, stool consistency will be assessed using the BSFS.
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose + Humiome® Post LB postbiotic on participant by Quality of Life score as assessed by IBS- QoL questionnaire | day 0, day 21, and day 42
  The quality of life will be assessed using the IBS-QOL scale. The participants will be asked to score based on their symptoms in the last month at day 0, day 21, and day 42.
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose + Humiome® Post LB postbiotic on participant by decreased Abdominal bloating as assessed by Gastrointestinal Quality of Life | day 0, day 21, and day 42
  The Gastrointestinal Quality of Life Index (GIQLI) is a validated 36-item tool for assessing health-related quality of life across five domains: core symptoms (10 items), physical (6 items), psychological (6 items), social (2 items), and disease-specific (8 items). Each item uses a 0-4 Likert scale, with higher scores indicating better quality of life. Total scores range from 0 to 144, where higher scores reflect improved quality of life.
To assess the efficacy on Increased percentage of responders to the treatment based on improvement on primary objective. The IBS-SSS is responsive to treatment; therefore, it has been used as a valid tool for performing responder analysis in IBS studies. | day 0, day 21 and day 42
  The number of responders will be calculated separately for the two definitions given below in the present study:
  1. 50 points change in IBS-SSS total score from baseline.
  2. 95 points change in IBS-SSS total score from baseline.
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on daily number of stool sample | Daily from start of the study to Week 6
  Will be assessed by Reduced Daily number of stools (stool frequency, assessed per IBS sub-type
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on Absolute difference in rescue medication consumption in active and placebo groups. | Daily from start of the study to Week 6
  Reduced Absolute difference in rescue medication consumption
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on Subjective global assessment of IP tolerability by participants. | Daily from start of the study to Week 6
  Will be measured by subjective global assessment of IP tolerability by participants
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on IBS-related mental stress relief | Day 0 and day 42
  Will be measured by Perceived stress scale (PSS)
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB on Gut Permeability assessment (Lactulose to Mannitol ratio test) [to be conducted in 30 participants in each arm] | Day 0 and day 42
  Will be measured by measuring the decrease in Lactulose Mannitol ratio (30 Participants per arm)
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on Stool pH & redox [to be conducted in 30 participants in each arm] | Day 0 and day 42
  Improved Stool pH (5.5 to 7.0) & decreased redox potential of stool [to be conducted in those participants who are undergoing LMR in each arm

OTHER OUTCOMES:
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on gut microbiome composition compared to baseline, each other and placebo | day 0 and day 42
  Improved Microbiome composition (i.e., increased in beneficial bifidobacteria) (on a selection of samples) will be analyzed using full shotgun sequencing (Illumina Hiseq 150 x2). This will be done on selection of samples
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on microbiome diversity compared to baseline, each other and placebo | day 0 and day 42
  Improved microbiome diversity (alpha and beta) will be analyzed (on a selection of samples) using full shotgun sequencing (Illumina Hiseq 150 x2) This will be done on selection of samples
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on fecal metabolomics profile compared to baseline, each other and placebo | day 0 and day 42
  Other fecal metabolites will be analysed for improvement (on a selection of samples) by an untargeted metabolomics approach using (semi-polar LC-MS/MS method. This will be done on selection of samples
To assess the efficacy of 6 weeks of daily consumption of two different mixes of HMO 2'-O-fucosyllactose (HMO-2FL) + Humiome® Post LB postbiotic (postbiotic-LB); on Changes in organic acids in fecal samples compared to baseline, each other and placebo | day 0 and day 42
  Improvement in fecal organic acids (acetate, propionate, butyrate, valerate, lactate) as analyzed (on a selection of samples) by a targeted quantitative SCFA method (GC-MS). This will be done on selection of samples

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Sadaghian, PhD, Study Director — DSM Nutritional Products, Inc.
Locations (12):
- India (12):
  - Shri. B. M. PatilMedical College,Hospital andResearch Centre, Vijayapura, Karnataka
  - Shivam Hospital, Dombivali, Maharashtra
  - Aster Aadhar Hospital, Kolhāpur, Maharashtra
  - D Y Patil, Navi Mumbai, Maharashtra
  - Dhanwantari Hospital, Pune, Maharashtra
  - Silver Birch, Pune, Maharashtra
  - Vishwaraj hospital, Pune, Maharashtra
  - D Y Patil Hospital, Medical college and research centre, Thane, Maharashtra
  - Dr. Naresh Bansal's Gastro & Liver Clinic, New Delhi, National Capital Territory of Delhi
  - Jaipur National University Institute of Medical Sciences and Research Centre, Jaipur, Rajasthan
  - Samvedna Hospital, New Colony, Ravindrapuri Varanasi
  - Gleneagles Global Hospitals, Hyderabad, Telangana